CLINICAL TRIAL: NCT03218852
Title: An Extended Follow-up of the Prospective Randomized, Controlled, Open-labeled Trial of Prednisone Plus Cyclophosphamide in Patients With Advanced Stage IgA Nephropathy
Brief Title: Extended Follow-up of Treatment of Prednisone Plus Cyclophosphamide in Patients With Advanced-stage IgA Nephropathy
Acronym: e-TOPplus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Shi, Clinical Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GGH2012-36-1
Record Dates: First submitted 2016-12-07; First posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Prednisone; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prednisone and cyclophosphamide (Experimental): 1. prednisone(0.5mg/kg/day*6 months)
  2. cyclophosphamide(1g intravenous use,per 1 month*6months);
  3. supportive care,including ACE-I or ARBs and blood pressure control
  Interventions: Drug: prednisone and cyclophosphamide
- prednisone alone (Experimental): 1. prednisone(0.5mg/kg/day*6months);
  2. supportive care,including ACE-I or ARBs and blood pressure control
  Interventions: Drug: prednisone alone

INTERVENTIONS:
Drug: prednisone and cyclophosphamide — Prednisone and cyclophosphamide are both administered to participants in this group.
  Arms: prednisone and cyclophosphamide
Drug: prednisone alone — Prednisone is administered to participants in this group.
  Arms: prednisone alone

SUMMARY:
This study is an extended follow-up of the study (ClinicalTrials.gov ID: NCT01758120)-Treatment of prednisone plus cyclophosphamide may be superior to treatment of prednisone alone in patients with advanced-stage IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven primary IgA nephropathy
* 18-70 years old
* elevated serum Creatinine and less than 3.0mg/dl
* with a written consent from participants to receive prednisone and/or cyclophosphamide

Exclusion Criteria:

* diabetes;
* contraindications for the treatment of prednisone and/or cyclophosphamide
* any treatment with steroids or immunosuppressive drugs prior to this study
* acute deterioration of renal function(including those of glomerular origin)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-12; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
the changes of kidney function or death | a total of 5 years of followup (addition of 2-year-follow up to the ClinicalTrial of NCT01758120)
  1. addition of 2-year-follow up to the ClinicalTrials.gov ID: NCT01758120;Time Frame:4 years and 5 years after the initiation of treatment
  2. the changes of estimated glomerular filtration rate (eGFR) or a combination of reaching end-stage renal disease (ESRD) or doubling of serum Creatinine or death

SECONDARY OUTCOMES:
the changes of proteinuria | a total of 5 years of followup (addition of 2-year-follow up to the ClinicalTrial of NCT01758120)
  1. addition of 2-year-follow up to the ClinicalTrials.gov ID: NCT01758120;Time Frame:4 years and 5 years after the initiation of treatment
  2. the changes of proteinuria
Number of Participants with Adverse Events | a total of 5 years of followup (addition of 2-year-follow up to the ClinicalTrial of NCT01758120)
  1. addition of 2-year-follow up to the ClinicalTrials.gov ID: NCT01758120;Time Frame:4 years and 5 years after the initiation of treatment
  2. Number of Participants with Adverse Events; adverse events include hair loss, vomiting, diarrhea, jaundice, leukopenia, anemia, thrombocytopenia, infections, allergic reactions and hemorrhagic cystitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No